CLINICAL TRIAL: NCT03940560
Title: Mesh Suture for Internal Load Bearing Closures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No clinical need to perform study
Sponsor: Wigmore Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-04-28; First posted 2019-05-07 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Suture; Complications, Mechanical; Suture; Complications, Infection or Inflammation; Suture, Complication
Keywords: suture; suture pull-through; suture sinus
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Intervention Model Description: Safety and efficacy study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Duramesh Suturable Mesh (Experimental): Use of Duramesh Suturable Mesh for internal load bearing closures
  Interventions: Device: Duramesh Suturable Mesh

INTERVENTIONS:
Device: Duramesh Suturable Mesh — Use of Duramesh Suturable Mesh for internal load bearing closures

SUMMARY:
Determine whether Mesh Suture achieves an acceptable safety and efficacy profile in load bearing internal tissue approximations. Mesh Suture has a novel design that permits tissue ingrowth and limits suture pull-through--items important for internal high-tension repairs

DETAILED DESCRIPTION:
Sutures are flexible linear elements that appose tissues and are "self-holding" with a surgically created knot. When tissues are under tension, such as the closure of an abdominal wall after laparotomy, the sutures cut through the tissues in what is known as "suture pull-through" and create incisional hernias. The hernia rate after primary laparotomy depends on the patient population, but is over 10%. In some high-risk populations, even with a small 3 cm laparoscopy incision, the hernia rate is over 30%. In primary hernia repair, use of sutures alone yields a 60% hernia recurrence rate at 10 years. Mesh has become commonplace in order to decrease incisional hernia recurrence rates in primary hernia repairs.

A novel mesh suture, designed at Northwestern University (Chicago, IL) by Dr. Gregory Dumanian, has shown improved outcomes in pre-clinical animal models and these results are included at the end of this document. Dr. Dumanian has employed the concept of using a mesh-like suture already in his clinical practice. He has cut strips from an FDA-approved piece of hernia mesh, and used them as sutures, tying them with knots.

Based on improved outcomes in pre-clinical and analogous clinical data in comparison to standard suture, Dr. Dumanian now proposes the use of a medical grade mesh suture of his design and fabrication in the load bearing internal tissue approximations. These are internal permanent sutures and will not be removed. They are made of the identical material (polypropylene) used in standard sutures.

Mesh Sutures are larger than standard sutures and they automatically flatten to help resist suture pull-through. Tissue ingrowth around the filaments and into the suture improves their hold.

ELIGIBILITY:
Inclusion Criteria:

* Deep orthopedic soft tissue approximation

Exclusion Criteria:

* Pregnancy
* Age less than 1 year old
* Repair of skin or other epithelial surfaces
* Poor subcutaneous tissues
* Ongoing infection

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgery healing complication, acute | 30 days
  Number of patients with infection, drainage, seroma, wound disruption over the mesh suture closure

SECONDARY OUTCOMES:
Surgery healing complication, delayed | Within 12 months
  Number of patients with infection, drainage, seroma, wound disruption, sinus over the mesh suture closure

CONTACTS AND LOCATIONS:
Overall Officials: Garen Koloyan, MD PhD, Principal Investigator — Wigmore Clinic
Locations (1):
- Wigmore Clinic, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03940560/Prot_000.pdf